CLINICAL TRIAL: NCT07108088
Title: Evaluation of the NEUROSWING Orthosis on Walking Speed in a Population With Dorsal and/or Plantar Flexor Deficits, With a View to a Reimbursement Application. Clinical Investigation: NS-BOOSST
Brief Title: Evaluation of the NEUROSWING Orthosis on Walking Speed in a Population With Dorsal and/or Plantar Flexor Deficits, With a View to a Reimbursement Application
Acronym: NS-BOOSST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ÖSSUR France (Industry)
Collaborators: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-A00585-44
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Multiple Sclerosis; Cerebral Palsy; Neuromuscular Deficits
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition A (Active Comparator): Condition A corresponds to the control phase where the patient will use the control device during 14 days.
  Interventions: Device: Carbon orthosis (control)
- Condition B (Experimental): Condition B corresponds to the experimental phase where the patient will use the experimental device during 14 days.
  Interventions: Device: NEUROSWING Orthosis (experimental) : carbon orthosis with an active ankle articulation

INTERVENTIONS:
Device: NEUROSWING Orthosis (experimental) : carbon orthosis with an active ankle articulation — The patients will use the experimental device during 14 days straight as well, then a washout period of 7 days with no interventons and then the comparator during 14 days straight. The order in which they will use each device will depend on the groupe they have been randomized in :
  * Arm 1 : Control device during 14 days, followed by a 7 day washout period, then exerimental device during 14 days
  * Arm 2 : Experimental device during 14 days, followed by a 7 day washout period, then control device during 14 days
  Arms: Condition B
Device: Carbon orthosis (control) — The patients will use the experimental device during 14 days straight as well, then a washout period of 7 days with no interventons and then the comparator during 14 days straight. The order in which they will use each device will depend on the groupe they have been randomized in :
  * Arm 1 : Control device during 14 days, followed by a 7 day washout period, then exerimental device during 14 days
  * Arm 2 : Experimental device during 14 days, followed by a 7 day washout period, then control device during 14 days
  Arms: Condition A

SUMMARY:
The aim of this randomized, cross-over, multi-center, intention-to-treat, open-label study study is to determine the benefits of the NEUROSWING device on gait speed in patients with dorsal and/or plantar flexor deficits, compared with the use of a carbon orthosis. Each patient will benefit in random order from a 14-day investigation period with the NEUROSWING device and a 14-day control period with a carbon orthosis. These two 2-week periods will be separated by one week, during which no orthosis will be worn and no evaluation will be carried out. Patients will be randomized to determine which phase they will start with. The primary endpoint is walking speed, which will be measured by comparing the results of the 10-meter walk test. For the secondary endpoints, patients will be assessed using the Functional Gait Assessment (FGA), the 6-minute test and an analysis system that will analyze other gait parameters (duration of the different phases of the gait cycle, cadence and step length). In order to carry out the assessments, each patient included will have 12 visits spread over 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Deficit of the dorsal and/or plantar flexors with at least one of the following components specific to the indication of an AFO:

  * steppage
  * foot drop,
  * spasticity,
  * failure to transfer weight-bearing,
  * instability of weight-bearing phase
  * compensatory hyperextension of the knee
  * Muscular deficiency of the dorsal and/or plantar flexors principal or accessory
* Ambulation possible with or without technical aids
* First time using an orthosis used in the study
* Being followed in one of the investigating centers whose management and rehabilitation in line with the study's visit schedule.
* Having freely consented to participate
* Affiliated with a social security scheme

Exclusion Criteria:

* Cognitive disorders, at the investigator's discretion, impacting the reliability of the clinical tests under study.
* Pathology in progressive phase at the time of inclusion that could significantly impact walking (e.g. MS, ALS, etc.) during the entire study period.
* Medically unstable (e.g. severe cardiovascular disorders) as judged by the investigating physician.
* Behavioral disorders (opposition, agitation, dementia) which, according to the investigator's judgment, would have an impact on walking.
* Already fitted with a carbon or NEUROSWING orthosis.
* Height over 214cm
* Weight over 193kg
* Pregnant, parturient or breast-feeding women
* Person deprived of liberty by a court order (including guardianship, curatorship and safeguard of justice) or administrative order
* Person under psychiatric care or admitted to a health or social establishment for purposes other than research
* Person in an emergency situation unable to give consent beforehand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Walking speed : 10m walk test | At all 12 visits from baseline (day 1), to end of study (day 35)

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | At baseline (day 1), day 14, day 22 and end of study (day 35)
  The Functional Gait Assessment (FGA) is a modification of the Dynamic Gait Index (DGI) that uses higher-level tasks to increase the applicability of the test to people with vestibular disorders and to eliminate the ceiling effect of the original test. Three items were added to the DGI because these were noted to be difficult in people with vestibular disorders.
  The FGA is used to assess postural stability during various walking tasks :
  * Gait on a Level Surface
  * Change in Gait Speed
  * Gait with Horizontal Head Turns
  * Gait with Vertical Head Turns
  * Gait and Pivot Turn
  * Step Over Obstacle
  * Gait with Narrow Base of Support
  * Gait with Eyes Closed
  * Ambulating Backwards
  * Steps
6 minute walk test | At baseline (day 1), day 14, day 22 and end of study (day 35)
Spatio-temoral gait analysis | At baseline (day 1), day 14, day 22 and end of study (day 35)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Leblong, Principal Investigator — Fondation Saint Helier
Locations (2):
- France (2):
  - IMPR du Bois de Lébisey, Hérouville-Saint-Clair
  - CMPR Bel-Air, La Membrolle-sur-Choisille